CLINICAL TRIAL: NCT01388660
Title: A Randomized, Open-label, Single-dose, Two-sequence, Two-period Crossover Study to Investigate The Pharmacokinetics Between a Tablet Containing 75 mg of Clopidogrel and 100 mg of Aspirin and The Simultaneous Administration of The Separate Formulations of The Two Drugs in Healthy Male Volunteers
Brief Title: Pharmacokinetic Assessment of Simultaneous Administration of Clopidogrel and Aspirin
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Doo-Yeoun Cho, Assitant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BCA006
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
Keywords: Healthy; Platelet Aggregation Inhibitors; Pharmacokinetics
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cloas (Experimental): A tablet containing 75 mg of Clopidogrel and 100 mg of Aspirin
  Interventions: Drug: Cloas
- Plavix/Astrix (Active Comparator): Simultaneous Administration of Plavix (75 mg of Clopidogrel) and Astrix (100 mg of Aspirin)
  Interventions: Drug: Plavix/Astrix

INTERVENTIONS:
Drug: Cloas — A tablet containing 75 mg of Clopidogrel and 100 mg of Aspirin, PO, 2 tablet once daily for Period I & II Day 1 (crossover manner)
  Arms: Cloas
Drug: Plavix/Astrix — Simultaneous Administration of Plavix (75 mg of Clopidogrel) and Astrix (100 mg of Aspirin), 2 tablets once daily for Period I & II Day 1 (crossover manner)
  Arms: Plavix/Astrix

SUMMARY:
This is a randomized, open-label, single-dose, two-sequence, two-period crossover study to investigate the pharmacokinetics between a tablet containing 75 mg of Clopidogrel and 100 mg of Aspirin and the simultaneous administration of the separate formulations of the two drugs in healthy male volunteers.

DETAILED DESCRIPTION:
Eligibility for participation of this study will be determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 4 weeks before study drug administration. Subjects suitable for this study will be admitted to the Clinical Trial Center of Ajou Medical Center on the day before dosing, and they will overnight-fasted from 10 p.m. of Day -1.

Subjects will be dosed study drug (a tablet containing 75 mg of Clopidogrel and 100 mg of Aspirin, or the simultaneous administration of the separate formulations of the two drugs) orally with 240 mL of water around 8 a.m. of Day 1. Subjects will be performed scheduled pharmacokinetic sampling upto 24 hours.

After 2 weeks of washout period, Subjects will be dosed study drug by crossover manner, and will be performed scheduled pharmacokinetic sampling upto 24 hours.

Study participation will be ended on post-study visit (Day 25).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 20 - 45 years
* With in 20% of ideal body weight, {Ideal body weight=[height(cm)-100]*0.9}
* Agreement with written informed consent

Exclusion Criteria:

* Clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal disease or mental disorder (Past history or present)
* Subject with symptoms of acute disease within 28 days of starting administration of investigational drug
* Subject with known for history which affect on the ADME of drug Clinically significant active chronic disease
* Inadequate result of laboratory test (especially, Platelet count < 150,000, Platelet count > 350,000, AST/ALT > 1.25 x UNL, Total bilirubin > 1.5 x UNL)
* Positive reaction in the HBs Ag, anti-HCV Ab, anti-HIV Ab, VDRL test
* Taking OTC(Over the counter)medicine including oriental medicine within 7 days
* Clinically significant allergic disease (Except for mild allergic rhinitis and dermatitis seems to be not need for medication)
* Subject with known for hypersensitivity reaction to clopidogrel or aspirin analog
* Not able to taking the institutional standard meal
* Previously make whole blood donation within 60 days or component blood donation within 30 days
* Previously participated in other trial within 90 days
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 30 g/day) and severe heavy smoker (cigarette > 1/2 pack per day)
* An impossible one who participates in clinical trial by investigator's decision including for reason of laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of Clopidogrel, Acetylsalicylic acid, and Salicylic acid | upto 24 hours after dosing
  Cmax (maximal plasma concentration) and AUC (area under the time-concentration curve) will be calculated from pharmacokinetic samplings

CONTACTS AND LOCATIONS:
Overall Officials: Doo-Yeoun Cho, MD, Principal Investigator — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea